CLINICAL TRIAL: NCT06343467
Title: Generic Volar Locking Plate Use in Distal Radius Fractures: A Prospective Randomized Study to Evaluate Clinical Outcomes and Cost Reduction
Brief Title: Do Generic Volar Locking Plates Provide Similar Outcomes at a Reduced Cost?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A17-376
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-03

CONDITIONS: Distal Radius Fractures
Keywords: Volar Locking Plate; Generic Implants
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Intervention Model Description: Surgeons alternated between using generic implants and conventional implants in their distal radius fracture patients over the course of six months.
Who Masked: Participant
Masking Description: Patients underwent the standard surgical consent, however the specific plate vendor that was used, was not specified by the physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Generic Implant (Experimental): Patients with an isolated distal radius fracture are treated surgically with a generic volar locking plate. All other surgical protocols remain unchanged.
  Interventions: Device: Generic Volar Locking Plate
- Conventional Implant (Active Comparator): Patients with an isolated distal radius fracture are treated surgically with a conventional, brand name volar locking plate of the surgeon's choice. All other surgical protocols remain unchanged.
  Interventions: Device: Conventional Volar Locking Plate

INTERVENTIONS:
Device: Generic Volar Locking Plate — Application of a generic volar locking plate is done in the generic implant arm compared to the other commonly used implants by surgeons in the conventional implant arm.
  Arms: Generic Implant
Device: Conventional Volar Locking Plate — Application of a conventional, brand name volar locking plate is done in the conventional implant arm compared to the generic implant arm.
  Arms: Conventional Implant

SUMMARY:
Across orthopedics, the investigators will be using the generic volar locking plates for patients undergoing open reduction and internal fixation (ORIF) of the distal radius using a block schedule, meaning one month we the generic implants and one month we use conventional implants from the surgeon's brand of choice. At the end of each month the health system will switch which type of implants (generic vs. conventional) they will use at their facilities. From a quality perspective each patient will be monitored both short and long term for complication and reoperation. This will be done through chart review.

DETAILED DESCRIPTION:
Patients will be consented to surgery per a standard surgical consent form. Six surgeons who regularly perform distal radius fracture (DRF) ORIF are included (five hand and one orthopaedic trauma fellowship-trained). Per the practice protocol, patients will either be treated with a generic plate or a brand name plate as described above. Ultimately, the decision to use a generic volar locking plate (VLP) is left up to surgeon discretion. All surgical and follow-up data will be collected. Implants used, age at time of surgery, weight, height, gender, race, ethnicity, comorbidities (diabetes, heart disease, etc.), complications including, but not limited to: readmission, reoperation, non-union, wound dehiscence, and lab tests will be collected. This will be evaluated all within 90 days following surgery. Implants will be cross referenced with the institution's data base to determine cost. All data will be collected on a secure server and be kept password protected. The primary outcome was 90-day postoperative complications (readmissions, reoperations, and mortality rates) by implant vendor type (generic vs. conventional). Secondary outcomes consisted of implant costs, estimated blood loss, and tourniquet time. An a priori power analysis was conducted to estimate the minimum sample size needed to adequately detect a difference in reoperation rates with a large effect size (Cohen's d=0.8). At a Type I error rate of 0.05, a power of 80%, and a 1:1 group allocation, the estimated sample size was 36 patients (18 generic VLPs vs. 18 conventional VLPs). Statistical significance was set to p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Isolated distal radius fracture
* Treated surgically with a volar locking plate

Exclusion Criteria:

* Volar locking plate not used
* Additional fixation was used
* Polytrauma (non-isolated injury)
* Open fracture
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Cunningham, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
This data will remain confidential and de-identified on our institution's servers.

REFERENCES:
- [Background] Walker JA, Althausen PL. Surgeon Attitudes Regarding the Use of Generic Implants: An OTA Survey Study. J Orthop Trauma. 2016 Dec;30 Suppl 5:S27-S31. doi: 10.1097/BOT.0000000000000722. PMID 27870671
- [Background] Waldrop VH, Laverty DC, Bozic KJ. Value-based Healthcare: Increasing Value by Reducing Implant-related Health Care Costs. Clin Orthop Relat Res. 2019 Feb;477(2):281-283. doi: 10.1097/01.blo.0000534683.24250.9c. No abstract available. PMID 29762154
- [Background] Miner HR, Slover JD, Koenig KM. Price Transparency and Consumer Perceptions of Generic and Brand-name Implants in Orthopaedic Surgery. Arch Bone Jt Surg. 2022 Sep;10(9):791-797. doi: 10.22038/ABJS.2022.51855.2558. PMID 36246025
- [Background] Mcphillamy A, Gurnea TP, Moody AE, Kurnik CG, Lu M. The Clinical and Economic Impact of Generic Locking Plate Utilization at a Level II Trauma Center. J Orthop Trauma. 2016 Dec;30 Suppl 5:S32-S36. doi: 10.1097/BOT.0000000000000721. PMID 27870672
- [Background] Khoo KM, Kim GW, Lindvall EM, Martirosian AK. Outcomes and Cost Comparison Between Generic and Conventional Cephalomedullary Nails in the Treatment of Peritrochanteric Femur Fractures. J Am Acad Orthop Surg. 2022 Feb 1;30(3):119-124. doi: 10.5435/JAAOS-D-21-00024. PMID 34715691
- [Background] Doxey SA, Huyke-Hernandez FA, Robb JL, Bohn DC, Cunningham BP. A Case Series of Surgically Treated Distal Radius Fractures: Implant Costs and Their Effect on Patient Outcomes. J Am Acad Orthop Surg Glob Res Rev. 2023 Jul 7;7(7):e23.00026. doi: 10.5435/JAAOSGlobal-D-23-00026. eCollection 2023 Jul 1. PMID 37428150
- [Background] Doxey SA, Huyke-Hernandez FA, Robb JL, Bohn DC, Cunningham BP. Implant cost variation in surgically treated distal radius fractures. J Orthop. 2023 Apr 7;39:45-49. doi: 10.1016/j.jor.2023.04.003. eCollection 2023 May. PMID 37125012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Detailed physical examination of patient with radiographic evaluation of distal radius fracture and indication for volar locking plate open reduction and internal fixation. Patients with open fracture observed on physical examination, polytrauma (any other fracture or medical instability), metaphyseal extension of the fracture, age less than 18 years, and fracture pattern not suitable for fixation with volar locking plate were excluded before assignment to groups.
Period: Overall Study
Arm/Group | Generic Implant | Conventional Implant
Started | 19 | 47
Completed | 19 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Implant | Conventional Implant | Total
Number analyzed (Participants) | 19 | 47 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 27 | 40
  >=65 years | 6 | 20 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.75 (12.16) | 60.74 (11.37) | 61.03 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 43 | 61
  Male | 1 | 4 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 47 | 66

OUTCOME MEASURES:

1. Primary Outcome: 90-day Reoperation Rate
Description: Reoperation for any reason postoperatively within 90 days after the date of surgery.
Time Frame: Within 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Implant | Conventional Implant
Number analyzed (Participants) | 19 | 47
Participants | 0 | 0

2. Primary Outcome: 90-day Readmission Rate
Description: Readmission to the hospital for any reason postoperatively within 90 days after the date of surgery.
Time Frame: Within 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Implant | Conventional Implant
Number analyzed (Participants) | 19 | 47
Participants | 0 | 0

3. Primary Outcome: 90-day Mortality Rate
Description: Patient death at any point within 90 days after the date of surgery.
Time Frame: Within 90 days postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Generic Implant | Conventional Implant
Number analyzed (Participants) | 19 | 47
Participants | 0 | 0

4. Secondary Outcome: Implant Cost
Description: The total cost of implants used in the procedure, including screws, pegs, volar locking plates, and disposable implants.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: United States Dollars
Arm/Group | Generic Implant | Conventional Implant
Number analyzed (Participants) | 19 | 47
United States Dollars | 702.38 (47.83) | 1348.61 (100.77)

5. Secondary Outcome: Tourniquet Time
Description: The total time in minutes from tourniquet inflation to deflation for a surgical case.
Time Frame: From tourniquet inflation to deflation during the procedure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Generic Implant | Conventional Implant
Number analyzed (Participants) | 19 | 47
minutes | 49.05 (19.2) | 45.06 (12.84)

6. Secondary Outcome: Estimated Blood Loss
Description: Estimated blood loss for the surgical case as reported by the surgeon in milliliters.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Generic Implant | Conventional Implant
Number analyzed (Participants) | 19 | 47
milliliters | 13.3 (10.2) | 13.2 (6.8)

ADVERSE EVENTS:
Time Frame: 90 days postoperatively
Arm/Group | Generic Implant | Conventional Implant
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/47
Other Adverse Events (participants affected / at risk) | 0/19 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT06343467/Prot_SAP_000.pdf